CLINICAL TRIAL: NCT00009971
Title: Phase II Trial Of Fenretinide (NSC-374551; IND-40, 294) In Patients With Relapsed Small Cell Lung Cancer
Brief Title: Fenretinide in Treating Patients With Recurrent Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068428; CCUM-9940; NCI-T99-0112
Record Dates: First submitted 2001-02-02; First posted 2003-01-27 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2003-10

CONDITIONS: Lung Cancer
Keywords: limited stage small cell lung cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Small Cell Lung Carcinoma | interventions — Fenretinide

ARMS (1):
- Arm I (Experimental): Patients receive oral fenretinide twice daily on days 1-7. Treatment continues every 21 days for at least 2 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: fenretinide

INTERVENTIONS:
Drug: fenretinide

SUMMARY:
Phase II trial to study the effectiveness of fenretinide in treating patients who have recurrent small cell lung cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the efficacy of fenretinide, in terms of complete and partial response rates, duration of response, and survival, in patients with recurrent small cell lung cancer.

II. Determine the toxicity of this regimen in these patients. III. Correlate the induction of apoptosis or the expression of molecular mediators of apoptosis in tumor cells with response rates, response duration, and survival in patients treated with this regimen.

OUTLINE: This is an open-label, multicenter study.

Patients receive oral fenretinide twice daily on days 1-7. Treatment continues every 21 days for at least 2 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed at 1 month.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed recurrent small cell lung cancer (SCLC) after platinum-containing chemotherapy regimen with or without thoracic radiotherapy

  * Limited stage or extensive stage SCLC
* Measurable disease

  * At least 20 mm by conventional techniques OR
  * At least 10 mm with spiral CT scan
* No pleural effusions, bone metastases, brain metastases, or abnormal radionucleotide scans as sole evidence of disease
* No symptomatic or uncontrolled brain or leptomeningeal disease

  * Previously treated brain metastases allowed if neurologically stable

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Zubrod 0-2

Hematopoietic:

* WBC at least 2,500/mm^3
* Platelet count at least 70,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 2 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No symptomatic heart disease
* No myocardial infarction within the past 6 months

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for 1 month before, during, and for 2 months after study
* No pre-existing retinal degenerative disease (e.g., retinitis pigmentosa or associated disorders)
* No other serious concurrent illness
* No other malignancy within the past 5 years except localized nonmelanoma skin cancer or carcinoma in situ

PRIOR CONCURRENT THERAPY:

Chemotherapy:

* At least 3 weeks since prior chemotherapy
* No more than 2 prior chemotherapy regimens

Endocrine therapy:

* Concurrent steroids allowed at stable dose

Radiotherapy:

* No prior radiotherapy to study lesions

Other:

* At least 3 weeks since prior systemic retinoid or carotenoid therapy
* No concurrent anticonvulsants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2000-11; Primary Completion 2005-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory P. Kalemkerian, MD, Study Chair — University of Michigan Rogel Cancer Center
Locations (2):
- United States (2):
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan